CLINICAL TRIAL: NCT01880554
Title: Clinical Utility of Contrast-enhanced Intraoperative Ultrasound in Surgery of Colorectal Liver Metastases. Phase II Clinical Trial.
Brief Title: Ultrasound Liver Intraoperative Imaging With SonoVue®
Acronym: ULIIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Bergonié (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IB2010-29
Record Dates: First submitted 2012-11-05; First posted 2013-06-19 (Estimated); Results first posted 2021-05-18 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2021-04

CONDITIONS: Liver Metastases From Colorectal Primary Cancer
Keywords: Liver metastases; Colorectal primary cancer; Contrast-enhanced ultrasound; Sonovue®

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Contrast-enhanced intraoperative ultrasound (Other): Contrast-enhanced intraoperative ultrasound
  Interventions: Device: Contrast-enhanced intraoperative ultrasound

INTERVENTIONS:
Device: Contrast-enhanced intraoperative ultrasound — Once the patient is included in the study, a staging procedure is performed in three stages before hepatic metastases treatment:
  Step # 1 preoperative (maximum 8 weeks before surgery Steps # 2 and # 3 intraoperative performed by the same surgeon in 2 stages

SUMMARY:
Hypothesis: Use of contrast ultrasound showed interesting results, which can increase ultrasonography sensitivity performed during surgery in the evaluation of operable liver metastases.

This study is a two-stage phase II multicenter study (Simon's two-stage).

DETAILED DESCRIPTION:
Hypothesis: Use of contrast ultrasound showed interesting results, which can increase ultrasonography sensitivity performed during surgery in the evaluation of operable liver metastases.

This study is a two-stage phase II multicenter study (Simon's two-stage).

ELIGIBILITY:
Inclusion Criteria:

1. Patient with histological proven colorectal cancer.
2. Operable liver metastases according to preoperative imagery. Operability is the possibility of treatment by resection and/or local destruction (radiofrequency, cryotherapy…).
3. Patient treated or not with preoperative chemotherapy.
4. With or without extra-hepatic metastases
5. Age ≥ 18 years.
6. Radiological assessment by CT and MRI liver and positron emission tomography scan (PETscan) within six weeks before surgery.
7. Patient affiliated to the Social Security system.
8. Signed informed consent.

Exclusion Criteria:

1. Known hypersensitivity to sulfur hexafluoride or another component of SonoVue®.
2. Patients with recent acute coronary syndrome or suffering from unstable ischemic heart disease, especially: evolving myocardial infarction, unstable angina during the last 7 days, recent coronary intervention or another factor suggesting clinical instability, acute heart failure, class III or IV heart failure, severe arrhythmias.
3. Patients with right-to-left shunt, severe pulmonary arterial hypertension, uncontrolled systemic hypertension, as patients suffering from respiratory distress syndrome.
4. Pregnant and lactating women.
5. Patients with contraindication for a CT scan, a MRI or a positron emission tomography (PET) with contrast.
6. Patients with indication of two step liver surgery.
7. Patients already included in the study.
8. Patient who couldn't be treated or followed up according to study criteria for psychological, social, family or geographical reasons. Patient deprived of liberty or under guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2011-06; Primary Completion 2016-09 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: EVRARD Serge, PU-PH, Study Chair — Institut Bergonié
Locations (1):
- Institut Bergonié, Bordeaux, Aquitaine, France

REFERENCES:
- [Background] Desolneux G, Isambert M, Mathoulin-Pelissier S, Dupre A, Rivoire M, Cattena V, Palussiere J, Dinart D, Bellera C, Evrard S. Contrast-enhanced intra-operative ultrasound as a clinical decision making tool during surgery for colorectal liver metastases: The ULIIS study. Eur J Surg Oncol. 2019 Jul;45(7):1212-1218. doi: 10.1016/j.ejso.2019.03.002. Epub 2019 Mar 10. PMID 30879929

RESULTS

PARTICIPANT FLOW:
Groups:
- Contrast-enhanced Intraoperative Ultrasound: Contrast-enhanced intraoperative ultrasound
  Contrast-enhanced intraoperative ultrasound: Once the patient is included in the study, a staging procedure is performed in three stages before hepatic metastases treatment:
  Step # 1 preoperative (maximum 8 weeks before surgery Steps # 2 and # 3 intraoperative performed by the same surgeon in 2 stages
Period: Overall Study
Arm/Group | Contrast-enhanced Intraoperative Ultrasound
Started | 68 (Patients enrolled in the study)
Population Eligible | 58
Population Eligible and Assessable | 54
Completed | 52 (Patients eligible and assessable according to two-stage Simon's design (primary outcome))
Not Completed | 16
Not completed — Protocol Violation | 14
Not completed — Simon's design requirements | 2

BASELINE CHARACTERISTICS:
Arm/Group | Contrast-enhanced Intraoperative Ultrasound
Number analyzed (Participants) | 52
Age, Continuous [Median (Standard Deviation); unit: years] | 62.8 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 35
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Cancer localization [Count of Participants; unit: Participants]
  Right Colon | 11
  Left Colon | 22
  Transverse Colon | 2
  Rectum | 17
Liver metastases [Count of Participants; unit: Participants]
  Synchronous | 29
  Metachronous | 23

OUTCOME MEASURES:

1. Primary Outcome: Clinical Utility of Intraoperative Contrast Ultrasound in the Surgery of Colorectal Cancer Liver Metastases.
Description: The clinical utility will be evaluated in terms of justified modification of the surgical procedure following contrast-enhanced intra-operative ultrasound (CE-IOUS), compared to the surgical procedure following conventional intra-operative ultrasound. For each patient, we will consider CE-IOUS to be clinically useful:
  * if the surgical procedure envisaged at the end of the CE-IOUS is different from the surgical procedure envisaged at the end of the conventional ultrasound
  * and if the surgical procedure envisaged at the end of the CE-IOUS is justified We reported the percentage of patients for whom there was a modified and justified surgical gesture following CE-IOUS.
Time Frame: At time of surgery
Population: We used a 2-stage Simon's design with the following assumptions:
  * maximum tolerated futility rate: 5%,
  * expected minimum utility rate: 15%,
  * Type I error of 10%,
  * power of 85%. Thus, 52 eligible and evaluable patients were required (25 in the first stage). First stage: stop, if CE-IOUS is not deemed clinically useful for at least one patient (4.0%).
  Second stage: CE-IOUS clinically useful if the planned surgical procedure is modified and justified for 5 or more patients (9.6%).
Measure: Number (95% Confidence Interval); unit: percentage of patients
Groups:
- Contrast-enhanced Intraoperative Ultrasound: Contrast-enhanced intraoperative ultrasound
  Contrast-enhanced intraoperative ultrasound: Once the patient is included in the study, a staging procedure is performed in three stages before hepatic metastases treatment:
  Step # 1 preoperative (maximum 8 weeks before surgery Steps # 2 and # 3 intraoperative performed by the same surgeon in 2 stages. Step #2 intraoperative ultrasound and step #3 Contrast-enhanced intraoperative ultrasound
Arm/Group | Contrast-enhanced Intraoperative Ultrasound
Number analyzed (Participants) | 52
percentage of patients | 7.7 [3.2 to 18.6]

2. Secondary Outcome: Clinical Utility of CE-IOUS in Subgroup of Patients Who Received Preoperative Chemotherapy
Description: The primary endpoint will be assessed in the subgroup of patients who received preoperative chemotherapy. As for the primary outcome, the clinical utility is evaluated in terms of justified modification of the surgical gesture envisaged following CE-IOUS, compared to the surgical gesture envisaged following a conventional intraoperative ultrasound.
  We reported the percentage of patients for whom there was a modified and justified surgical gesture following CE-IOUS in the subgroup of patients who received preoperative chemotherapy.
Time Frame: at time of surgery
Population: Subgroup of patients with preoperative chemotherapy
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Contrast-enhanced Intraoperative Ultrasound
Number analyzed (Participants) | 41
percentage of patients | 7.31 [2.52 to 19.43]

3. Secondary Outcome: Performance Evaluation of Intraoperative Ultrasound Contrast: Detection Rate Per Lesion
Description: Detection of malignant lesions by CE-IOUS in chemotherapy-free patients within 3 post-operative months. The detection rate is defined as the proportion of malignant lesions for which there is concordance between the diagnosis established by CE-IOUS and the reference examination.
Time Frame: up to 3 months after surgery
Population: There were 22 (40.7%) out of 54 chemotherapy-free patients within 3 post-operative months
Measure: Number; unit: proportion of lesions
Arm/Group | Contrast-enhanced Intraoperative Ultrasound
Number analyzed (Participants) | 22
proportion of lesions | 0.75

4. Secondary Outcome: Description of Technical Arrangements for the CE-IOUS
Description: Description of technical arrangements for the CE-IOUS duration. The length of time during which contrast injection was useable.
Time Frame: At time of contrast-enhanced IOUS
Measure: Median (Full Range); unit: seconds
Arm/Group | Contrast-enhanced Intraoperative Ultrasound
Number analyzed (Participants) | 54
seconds | 225 [105 to 307]

5. Secondary Outcome: Performance Evaluation of Intraoperative Ultrasound Contrast Per Lesion: Characterisation Rate
Description: Characterisation rate for focal liver lesions: the proportion of lesions whose nature on CE-IOUS is identical to the nature of the lesions defined by the reference examinations among all the lesions seen on CE-IOUS (malignant and benign)
Time Frame: up to 3 months after surgery
Measure: Number; unit: proportion of lesions
Arm/Group | Contrast-enhanced Intraoperative Ultrasound
Number analyzed (Participants) | 54
proportion of lesions | 0.94

ADVERSE EVENTS:
Arm/Group | Contrast-enhanced Intraoperative Ultrasound
Serious Adverse Events (participants affected / at risk) | 11/54
Other Adverse Events (participants affected / at risk) | 2/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Contrast-enhanced Intraoperative Ultrasound (N=54)
Peritonitis (Infections and infestations) | 2
Hypertension (Vascular disorders) | 1
Eventration (Surgical and medical procedures) | 1
Biliary fistula (Hepatobiliary disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Bile collection secondary to a biliary tract wound (Hepatobiliary disorders) | 1
Fistule anastomose colorectale (Gastrointestinal disorders) | 1
Hepatic failure (Hepatobiliary disorders) | 1
Peri-hepatic Blood Collection (Vascular disorders) | 1
Stercoral peritonitis (Infections and infestations) | 1
Asthenia (General disorders) | 1
Right cry (Respiratory, thoracic and mediastinal disorders) | 1
Acute pancreatitis (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Contrast-enhanced Intraoperative Ultrasound (N=54)
Anemia (Blood and lymphatic system disorders) | 1
Hepatocellular insufficiency (Hepatobiliary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No